CLINICAL TRIAL: NCT06734260
Title: Optimization of Keverprazan-amoxicillin Dual Therapy for Eradicating Helicobacter Pylori Infection：a Multicenter, Prospective, Randomized Controlled Study
Brief Title: Optimization of Keverprazan-amoxicillin Dual Therapy for Eradicating Helicobacter Pylori Infection
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, chenhonglei, Doctor, Eighth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-229-02
Record Dates: First submitted 2024-12-12; First posted 2024-12-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Helicobacter Pylori Eradication Rate
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- H-KA-dual-14 (Active Comparator): 14 days(Keverprazan Hydrochloride tablets 20 mg/time, 2 times/day, oral
  +Amoxicillin 1000mg/ time, 3 times/day, oral)
  Interventions: Drug: Keverprazan Hydrochloride tablets + high dose amoxicillin
- L-KA-dual-14 (Experimental): 14 days(Keverprazan Hydrochloride tablets 20 mg/time, 2 times/day, oral
  +Amoxicillin 1000mg/ time, 2 times/day, oral)
  Interventions: Drug: Keverprazan Hydrochloride tablets + low dose amoxicillin
- H-KA-dual-10 (Experimental): 10 days(Keverprazan Hydrochloride tablets 20 mg/time, 2 times/day, oral
  +Amoxicillin 1000mg/ time, 3 times/day, oral)
  Interventions: Drug: Keverprazan Hydrochloride tablets + high dose amoxicillin（H-KA-10d）

INTERVENTIONS:
Drug: Keverprazan Hydrochloride tablets + high dose amoxicillin — Keverprazan Hydrochloride tablets 20 mg/time, 2 times/day, oral Amoxicillin 1000mg/ time, 3 times/day, oral, for 14 day
  Other Names: H-KA-14d
  Arms: H-KA-dual-14
Drug: Keverprazan Hydrochloride tablets + low dose amoxicillin — Keverprazan Hydrochloride tablets 20 mg/time, 2 times/day, oral Amoxicillin 1000mg/ time, 2 times/day, oral, for 14 day
  Other Names: L-KA-14d
  Arms: L-KA-dual-14
Drug: Keverprazan Hydrochloride tablets + high dose amoxicillin（H-KA-10d） — Keverprazan Hydrochloride tablets 20 mg/time, 2 times/day, oral Amoxicillin 1000mg/ time, 3 times/day, oral, for 10 day
  Other Names: H-KA-10d
  Arms: H-KA-dual-10

SUMMARY:
Eradication of HP can significantly improve and reduce HP-related diseases. A 10-14 day quadruple regimen containing bismuth as first-line treatment, achieving an eradication rate of more than 85%. However, some disadvantages of these quadruple regimens, such as severe adverse reactions, high medical costs and low compliance, prevent their application in clinical practice. High-dose proton pump inhibitors (PPI) combined with amoxicillin can be used as the first-line treatment for HP eradication, with good efficacy and compliance and low rate of adverse reactions. However, the acid inhibition effect of PPI mainly depends on the degree of individual metabolism of proton pump,which might influence the eradication effect. Keverprazan, a new competitive potassium acid blocker(P-CAB), is not affected by gene polymorphism, and has the advantage of stronger and longer inhibition effect on gastric acid compared with PPIs. This study aimed to evaluate two different doses of therapy (1 g b.i.d. vs. 1.0 g t.i.d.) and two different durations of therapy (14 vs.10 days) to gain insights of the effectiveness of Keverprazan-amoxicillin dual therapy .

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 75 years;
2. Adult subjects who voluntarily signed written informed consent approved by the ethics committee to consent to participate in this study before the start of any study procedure;
3. Subjects who can understand and comply with the protocol requirements and agree to attend all study visits;
4. During the screening phase, patients who were Hp positive and required Hp eradication therapy as judged by the investigator, and patients who had failed Hp eradication for the first time;
5. Participants agreed to use appropriate medical methods of contraception (except medically sterilized status) during the study.

Exclusion Criteria:

* 1. Participated in other clinical studies within 4 weeks before screening; 2. Pregnant or lactating women; 3. Known allergy to keverprazan, esomeprazole, penicillins or other beta-lactams, macrolide antibiotics, nitrofuran antibiotics, or bismuth (including any relevant adjuvants). If skin sensitivity testing (skin testing) was required, it was performed at visit 1 according to routine medical practice; 4. Participants had a history of drug (including but not limited to opioids) abuse or alcohol abuse (> 14 units of alcohol per week, 1 unit of alcohol ≈360mL of approximately 5% beer or 45 ml of approximately 40% spirits or 150 ml of approximately 12% wine) in the year before the screening visit; 5. The subjects had Zolie-Ellison syndrome, gastric acid hypersecretion, or a history of gastric acid hypersecretion; 6. The subject has undergone previous surgery or operation that may affect gastric acid secretion or drug absorption, such as subtotal gastrectomy, total gastrectomy, vagotomy, intestinal resection, etc. Simple surgery for perforation, appendectomy, cholecystectomy, and endoscopic resection of benign tumors are acceptable; 7. "Warning" symptoms such as odynophagia, severe dysphagia, bleeding, weight loss, anemia, or hematochezia that might indicate the presence of a malignant GI lesion, unless a malignant lesion was ruled out by endoscopy; 8. A history of malignancy within 5 years before screening (participants were allowed to participate if they had been cured of skin basal cell carcinoma or cervical carcinoma in situ); 9.. Upper gastrointestinal endoscopy showed acute upper gastrointestinal bleeding, active gastric or duodenal ulcer, acute gastric or duodenal mucosal injury; 10. According to the investigator's judgment, the subject has uncontrolled and unstable liver, kidney, cardiovascular, respiratory, gastrointestinal, endocrine, hematological, central nervous system or mental diseases, etc., and participating in the study may affect the safety of the subject or the interpretation of the study results; 11. Subjects who plan to be hospitalized for surgical treatment during the study; 12. H2-receptor antagonist or PPI use within 14 days prior to screening 13C-urea breath test; During the screening period, antibiotics, bismuth and some traditional Chinese medicine with antibacterial effect were taken within 28 days before 13C-urea breath test; 13. Abnormal laboratory test results at screening in any of the following: AST > upper limit of normal (ULN); ALT > Upper limit of normal (ULN); Total bilirubin > ULN; creatinine > 1.5 times ULN; 14. The subjects had clinically significant abnormal electrocardiogram (ECG), including severe arrhythmia, multifocal premature ventricular contractions (PVC), second degree or above atrioventricula

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 477 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
H. pylori eradication rate | 6 weeks
  Rate of h. pylori successfully eradicated；13C-urea breath testthat will be used to assess this outcome measure

SECONDARY OUTCOMES:
Adverse Event | 6 weeks
  Rate of adverse event, serious adverse event; Questionnaire that will be used to assess this outcome measure.
Medical financial burden | 6 weeks
  Medical financial burden；Questionnaire that will be used to assess this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Shanshan Wei, MD, Study Chair — The Eighth Affiliated Hospital,sun Yet-san University; Huizhen Xiong, Study Chair — The Eighth Affiliated Hospital,sun Yet-san University; Meifang Ye, Study Chair — The Eighth Affiliated Hospital,sun Yet-san University; Jianfeng Zhong, Study Chair — The Eighth Affiliated Hospital,sun Yet-san University; Wei Liu, Study Chair — The Eighth Affiliated Hospital,sun Yet-san University; Fang Liu, Study Chair — The Eighth Affiliated Hospital,sun Yet-san University; Ting Zhou, Study Chair — The Eighth Affiliated Hospital,sun Yet-san University; Qiucheng Li, Study Chair — The Eighth Affiliated Hospital,sun Yet-san University
Locations (4):
- China (4):
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Puning Overseas Chinese Hospital, Puning, Guangdong
  - Eighth Affiliated Hospital,Sun Yet-san University, Shenzhen, Guangdong
  - Xiangyang Hospital of Traditional Chinese Medicine, Xiangyang, Hubei

IPD SHARING:
Plan to Share IPD: No
The datasets used and analysed during the current study available from the corresponding author on reasonable request.